CLINICAL TRIAL: NCT00311610
Title: Phase II Trial of LE SN38 in Patients With Metastatic Colorectal Cancer After Progression on Oxaliplatin
Brief Title: Liposomal SN-38 in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-80402; U10CA031946 (NIH); CALGB-80402; CDR0000467234 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SN-38 liposome (Experimental): Patients receive SN-38 liposome IV over 90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  After completion of study treatment, patients are followed every 3 months for up to 3 years.
  Interventions: Drug: SN-38 liposome

INTERVENTIONS:
Drug: SN-38 liposome — 38 mg/sq m IV infusion over 30 min q 21 days (1 cycle) until progression

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposomal SN-38, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well liposomal SN-38 works in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate following treatment with SN-38 liposome as a second-line treatment in patients with metastatic colorectal cancer.

Secondary

* Determine the toxicity profile of this drug in these patients.
* Determine the proportion of patients treated with this drug who experience any grade 3 or greater toxicity.
* Determine progression-free survival and overall survival for patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive SN-38 liposome IV over 90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically determined metastatic colorectal cancer*

  * Primary lesion confirmed endoscopically, surgically, or radiologically NOTE: * Patients with a history of colorectal cancer treated by surgical resection who develop radiological or clinical evidence of metastatic cancer do not require separate histological or cytological confirmation of metastatic disease, unless more than 5 years between primary surgery and development of metastatic disease OR primary cancer was stage I
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan

  * Nonmeasurable lesions include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* UGT1A1*1 homozygous or UGT1A1*28 heterozygous genotype status

  * Patients with homozygous UGT1A1*28 genotype not eligible
* Received at least 1 prior regimen with oxaliplatin for metastatic disease
* Recurrent disease following prior adjuvant therapy allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine normal
* Bilirubin normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception duration and for 3 months after completion of study treatment
* No known Gilbert's disease or other chronic liver disease
* No colonic or small bowel disorders (e.g., inflammatory bowel disease, Crohn's disease, or ulcerative colitis) that predispose the patients to uncontrolled diarrhea (i.e., > 3 watery or soft stools daily at baseline in patients without a colostomy or ileostomy)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* No prior irinotecan
* Prior pelvic radiotherapy allowed as long as measurable lesion is outside irradiated field
* No concurrent palliative radiotherapy
* No other concurrent chemotherapy
* No concurrent steroids except those given for adrenal failure, hormones for non-disease-related conditions (e.g., insulin for diabetes), or intermittent dexamethasone as an antiemetic or for prevention of infusion reaction

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2007-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Objective response rate | q 2 cycles during tx

SECONDARY OUTCOMES:
Toxicity | q cycle during tx
Progression-free survival | 3 years
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Allyson Ocean, MD, Study Chair — Weill Medical College of Cornell University
Locations (10):
- United States (10):
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio

REFERENCES:
- [Result] Ocean AJ, Niedzwiecki D, Atkins JN, et al.: LE-SN38 for metastatic colorectal cancer after progression on oxaliplatin: results of CALGB 80402. [Abstract] J Clin Oncol 26 (Suppl 15): A-4109, 2008.